CLINICAL TRIAL: NCT07196800
Title: Effect of Dose Variations of High-Power Laser Therapy on Patients With Nonspecific Cervical Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Deraya University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: physio 2 2025
Record Dates: First submitted 2025-09-20; First posted 2025-09-29 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Neck Pain
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- lower dose laser therapy (Active Comparator)
  Interventions: Radiation: High intensity laser therapy (low dose) combined with conventional physiotherapy program
- higher dose laser therapy (Experimental)
  Interventions: Procedure: High intensity laser therapy (High dose) combined with conventional physiotherapy program

INTERVENTIONS:
Radiation: High intensity laser therapy (low dose) combined with conventional physiotherapy program — 840 joules delivered during each session combined with conventional physiotherapy program Participants
  Arms: lower dose laser therapy
Procedure: High intensity laser therapy (High dose) combined with conventional physiotherapy program — 2632 joules delivered during each session combined with conventional physiotherapy program
  Arms: higher dose laser therapy

SUMMARY:
Nonspecific neck pain, defined as pain without a specific underlying pathology, is a common musculoskeletal disorder that affects a significant proportion of the global population. Neck pain often results in considerable discomfort and functional limitations, impacting individuals' quality of life and ability to perform daily tasks. Estimates suggest that up to 30% of adults experience neck pain annually. The condition ranks among the top causes of disability worldwide, contributing to substantial personal and societal burdens, including lost work productivity and increased healthcare costs.

ELIGIBILITY:
Inclusion Criteria:

* unilateral or bilateral CNP
* Experiencing moderate to severe neck pain, defined as a Visual Analog
* Scale (VAS) score of ≥4.
* Cervical Range of Motion (ROM) Limitation: Documented restriction in cervical ROM compared to normal values for age and gender, to ensure the condition's impact on functional mobility
* Patients agreed not to take any medication(anti-inflammatories, analgesics, or muscle relaxants) throughout the course of the study or receive any type of treatment for neck pain

Exclusion Criteria:

* Previous Cervical Surgery: Patients with a history of cervical spine surgery will be excluded to eliminate potential influences from post-surgical changes on the outcomes
* Diagnosed with cervical disc prolapse as confirmed by clinical evaluation and imaging studies (MRI or CT scans).
* History of malignancy in the cervical region or other serious medical conditions.
* Severe comorbidities that may affect treatment outcomes (e.g., uncontrolled diabetes, cardiovascular diseases).
* Pregnancy or lactation.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-03-10 (Actual); Primary Completion 2025-11-10 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Pain assessment | 4 weeks
  where participants will rate their pain on a scale from 0 (no pain) to 10 (worst pain imaginable).
Cervical Range of Motion (ROM): | 4 weeks
  ROM will be measured using an OB goniometer in three planes

CONTACTS AND LOCATIONS:
Locations (1):
- Deraya university physiotherapy clinic, Minya, Egypt

IPD SHARING:
Plan to Share IPD: Undecided